CLINICAL TRIAL: NCT01615887
Title: Effects of Lisdexamfetamine on Bradyphrenia in Multiple Sclerosis
Brief Title: Study of Lisdexamfetamine Sulfate to Treat Cognitive Dysfunction in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Bianca Weinstock-Guttman, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU2570309B
Record Dates: First submitted 2011-03-23; First posted 2012-06-11 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- lisdexamfetamine sulfate (Experimental): 30mg lisdexamfetamine OD, increased to 70mg OD over 4 weeks and continued on 70mg OD for 4 weeks
  Interventions: Drug: lisdexamfetamine sulfate
- Sugar pill (Placebo Comparator): Placebo will be administered in the same fashion as the treatment arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lisdexamfetamine sulfate — 30mg lisdexamfetamine OD, increased to 70mg OD over 4 weeks and continued on 70mg OD for 4 weeks
  Other Names: Vyvanse
  Arms: lisdexamfetamine sulfate
Drug: placebo — sugar pill
  Arms: Sugar pill

SUMMARY:
Amphetamines have been shown to improve cognition but its use is limited due to its side effects. Lisdexamfetamine is an amphetamine pro-drug, minimizing these effects and has been safely used in children and adults with Attention Deficit Hyperactivity Disorder (ADHD). The investigators hypothesize that lisdexamfetamine may improve cognitive abilities in MS patients with documented cognitive dysfunction. Because lisdexamfetamine is a stimulant its positive effects should be observed primarily in the domains of processing speed and working memory. The investigators therefore propose a study in which the primary objective will be to assess the efficacy of lisdexamfetamine in improving attention and processing speed in MS. The secondary objectives will be (a) the assessment of the safety and tolerability of lisdexamfetamine in the MS population, and (b) to test for effects of the drug on other cognitive domains, depression, and self and informant reports of cognitive and executive function demanding activities and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Males/Females who are ≥ 18 years old and < 55 years old and are capable of understanding and complying with the protocol, including speaking and writing fluent English and having at least a 9th grade education.
* Have a diagnosis of either Relapsing Remitting or Secondary Progressive MS, as per revised McDonald's Criteria (68).
* Have not received steroids in last thirty (30) days or a relapse in the last ninety (90) days, and whose MS is considered stable.
* Presence of cognitive dysfunction characterized by slowed processing speed as indicated by a score of -1.5 SD below age/education matched norms on the SDMT or the PASAT.
* An Expanded Disability Status Scale (EDSS) of ≤ 6.5
* Have given written informed consent prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care.
* Are capable of performing the requirements of a NP test battery including at least 20/70 near visual acuity by near vision chart, with correction allowed.
* If female, must neither be pregnant nor breast-feeding and must either (a) be > 12 months post-menopausal or surgically sterilized, or (b) agree to use an acceptable method of birth control for the duration of the study. Abstinence will not be considered an acceptable method of birth control.

Exclusion Criteria:

* Have cognitive deficits caused by concomitant medication usage or other significant neurological/psychological disease e.g. Alzheimer's disease, Parkinson's disease, stroke, transient ischemic attack, Vascular Dementia, Huntington's disease, traumatic brain injury or chronic CNS infection
* Have evidence of other medical cause(s) of cognitive impairment
* Have evidence of major depression as determined by a positive BDIFS and clinician interview
* Have uncontrolled or labile hypertension, tachycardia, cardiovascular or cerebrovascular disease
* Have demonstrated a hypersensitivity to amphetamines in the past
* The following concomitant medications are not permitted to be used within 28 days of enrollment or during the study

  * Monoamine Oxidase Inhibitors
  * Inhaled Beta2-agonists
  * Sympathomimetics
  * Antipsychotic agents
  * Modafinil
  * Tricyclic Antidepressants
  * Anticonvulsants other than gabapentin and pregabalin
* The following medications are permitted if the patient has been on a stable dose for ≥ 6 weeks:

  * Short acting benzodiazepines, qhs administration only
  * Gabapentin and pregabalin Cholinesterase inhibitors other than donepezil, galantamine, and rivastigmine
  * Memantine
  * Anti-spasmodics
  * Selective serotonin reuptake inhibitors and serotonin-norepinephrine reuptake inhibitors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaleida Health, Jacobs Neurological Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Started | 41 | 22
Completed | 29 | 19
Not Completed | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill | Total
Number analyzed (Participants) | 29 | 19 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (8.0) | 46.7 (8.5) | 47.7 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 26 | 18 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 19 | 48

OUTCOME MEASURES:

1. Primary Outcome: Symbol Digit Modalities Test (SDMT)
Description: The Symbol Digit Modalities Test (SDMT) presents a series of nine symbols, each paired with a single digit in a key at the top of a stimulus page. Subjects voice the number associated with each symbol as rapidly as possible. The examiner records the total amount of responses completed. The task continues for 90 seconds with the research staff recording responses. The SDMT score ranges from 0 to 110, with higher values representing a better outcome in cognitive processing speed.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
score on a scale | 36.9 (8.7) | 46.8 (7.5)

2. Primary Outcome: Paced Auditory Serial Audition Test (PASAT)
Description: The PASAT is a test requiring attention and vigilance. In this test, the patient listens to a tape recording of digits presented one at a time. The task for the patient is to add each number to the one immediately preceding it. For example, the recording might present the numbers 1, 7, 5, 4. The patient adds the first two numbers (1 + 7) and responds with the number 8. The patient then adds the second two numbers (7 + 5) and responds with the number 12. The patient then adds the third two numbers (5 + 4) and responds with the number 9. This continues for a total of 61 numbers presented in a random order. The patients score is the total number correct out of 60 (Stebbins et al. 2007). The PASAT score ranges from 0 to 60, with higher values representing a better outcome in cognitive processing speed.
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
score on a scale | 32.0 (12.5) | 37.4 (12.1)

3. Secondary Outcome: California Verbal Learning Test - 2nd Edition
Description: The California Verbal Learning Test Second Edition (CVLT2) begins with the examiner reading a list of 16 words. Patients listen to the list and report as many of the items as possible. After recall is recorded, the entire list is read again. Altogether, there are five learning trials, the total correct of all trials is summed together creating a total verbal learning score. The CVLT-II total verbal learning score ranges from 0 to 80, with higher values representing a better outcome in verbal learning/memory.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
score on a scale | 44.9 (11.5) | 49.2 (10.2)

4. Secondary Outcome: Brief Visuospatial Memory Test - Revised
Description: The Brief Visuospatial Memory Test Revised (BVMTR) presents six abstract designs for 10 seconds. The display is removed from view and patients render the stimuli via pencil on paper manual responses. There are three learning trials in which patients attempt to replicate the stimuli previously presented. Patients are given a score for all three trials based on correct location and accuracy of the replicated stimuli. Each trial can be awarded up to 12 points, the sum of total points awarded across all three trials is the total learning score. The BVMT-R total learning score ranges from 0 to 36, with higher values representing a better outcome in visuospatial learning/memory.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
score on a scale | 15.2 (6.1) | 18.7 (5.5)

5. Secondary Outcome: Vitals
Description: Heart rate
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
beats/min | 72.3 (11.7) | 76.9 (10.6)

6. Secondary Outcome: Vitals (Diastolic Blood Pressure)
Description: diastolic blood pressure
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm hg (millimeters of mercury)
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
mm hg (millimeters of mercury) | 75.1 (11.3) | 77.7 (7.7)

7. Secondary Outcome: Vitals (Systolic Blood Pressure)
Description: systolic blood pressure
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mm hg (millimeters of mercury)
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Number analyzed (Participants) | 29 | 19
mm hg (millimeters of mercury) | 127.3 (15.9) | 121.6 (13.1)

ADVERSE EVENTS:
Time Frame: adverse events data were collected over the 8-week study period. During the first 4 weeks adverse event data was collected weekly and then once more 4 weeks later.
Description: Participants were monitored for serious adverse events weekly during the first 4 weeks and then once more 4 weeks later. During this time no serious adverse events were reported by subjects and no objective measures suggested any serious adverse events took place.
Arm/Group | Lisdexamfetamine Sulfate | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/22
Other Adverse Events (participants affected / at risk) | 23/41 | 12/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Sulfate (N=41) | Sugar Pill (N=22)
dry mouth (Gastrointestinal disorders) | 15 | 2
nausea (Gastrointestinal disorders) | 5 | 1
palpitations (Cardiac disorders) | 5 | 1 — subjective report of feeling palpitations
increased heart rate (Cardiac disorders) | 11 | 2 — increased by 15 or more beats per minute
Increased systolic blood pressure (Cardiac disorders) | 4 | 1
increased diastolic blood pressure (Cardiac disorders) | 8 | 1
flushing/feeling warm (Cardiac disorders) | 3 | 0
headache (General disorders) | 8 | 1
lightheadedness (General disorders) | 4 | 0
Paresthesias (General disorders) | 3 | 1
weight loss (Metabolism and nutrition disorders) | 3 | 0
decreased appetite (Metabolism and nutrition disorders) | 11 | 1
anxiety (Psychiatric disorders) | 5 | 0
agitation (Psychiatric disorders) | 3 | 0
mania (Psychiatric disorders) | 4 | 1
body aches and cramps (General disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No